CLINICAL TRIAL: NCT05321888
Title: Effects of Mechanical Ventilation With and Without Postural Drainage on Oxygen Saturation, Airway Clearance in Burn Patients With Acute Respiratory Distress Syndrome
Brief Title: Mechanical Ventilation With and Without Postural Drainage in Burn Patients With ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/220310
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Burns (Physical Finding)
Keywords: Respiration; Artifical Respiration; Postural drainage; Respiratory distress syndrome; Respiratory physiological phenomena
MeSH Terms: conditions — Burns; Respiratory Aspiration; Respiratory Distress Syndrome | interventions — Respiration, Artificial; Drainage, Postural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Ventilation (Active Comparator): Mechanical Ventilation
  Interventions: Other: Mechanical Ventilation
- Mechanical Ventilation with Postural drainage (Experimental): Mechanical Ventilation with Postural drainage
  Interventions: Other: Mechanical Ventilation with Postural drainage

INTERVENTIONS:
Other: Mechanical Ventilation — Standard Protocol
  Arms: Mechanical Ventilation
Other: Mechanical Ventilation with Postural drainage — This Group will be treated by postural drainage and mechanical ventilation for two consecutive days
  Arms: Mechanical Ventilation with Postural drainage

SUMMARY:
Inhalation injury become a more common cause of death in burn patients but alone the smoke injury has low mortality rate. It is reported that a combination of smoke injury with cutaneous burn increases the mortality rate and predispose to Acute Respiratory Distress Syndrome. This experimental study aims to report the benefits of postural drainage on the respiratory system in burn patients. This study will determine the effects of postural drainage on oxygen saturation, airway clearance in burn patients with Acute Respiratory Distress Syndrome by comparing mechanical ventilation with and without the application of postural drainage. A randomized clinical trial will be conducted in the data and will be collected from the ICU of Jinnah Burn & Reconstructive Surgery Centre and Shafique Aziz Free Burn Centre through consecutive sampling through technique on 50 patients which will be allocated through sealed opaque enveloped into Group A and Group B. Pre and post treatment value of oxygenation and other variables for both group will be recorded by using APACHE II. Group A will be treated by postural drainage and mechanical ventilation for two consecutive days. Similarly, Group B will be treated by mechanical ventilation only. Data will be analyzed using SPSS software 25. After assessing the normality of data by the Shapiro-Wilk test, it will be decided either parametric or non-parametric tests will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender male and female are included.
* Patient age should be between 10-40 years
* Patients that are on mechanical ventilation
* Patients with inhalation injury
* Patients undergo mechanical ventilation for >48 hours

Exclusion Criteria:

* Patient with no past medical history of Lung disease
* Subject with more than 80% of burn according to Rule of Nine
* Patients with cardiac instability such as recent Myocardial infarction, Unstable angina and severe hypotension and hypertension

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II | SECOND DAY
  APACHE stands for Acute Physiology and Chronic Health Evaluation II which is mostly used in the ICU to check the severity of the disease. This score measures the seriousness of sickness and the adequacy of clinical medical services and the doctor's decision allowing more exact prognostic delineation of seriously sick patients. APACHE II an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death The tool consists of twelve physiological variables. From which we are using five variables are age, Respiratory rate, Oxygenation (FiO2, PaO2), Mean Arterial Pressure, Glasgow comma score, Temperature, Systolic Blood Pressure, Heart Rate, Arterial pH, Acute Renal Failure, History of organ failure other than this Mechanical ventilation or CPAP, gender, and sputum profiles were also included which are not the part of this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Burn & Reconstructive Surgery Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva L, Garcia L, Oliveira B, Tanita M, Festti J, Cardoso L, Lavado L, Grion C. Acute respiratory distress syndrome in burn patients: incidence and risk factor analysis. Ann Burns Fire Disasters. 2016 Sep 30;29(3):178-182. PMID 28149245
- [Background] Chung F, Mueller D. Physical therapy management of ventilated patients with acute respiratory distress syndrome or severe acute lung injury. Physiother Can. 2011 Spring;63(2):191-8. doi: 10.3138/ptc.2010-10. Epub 2011 Apr 13. No abstract available. PMID 22379259
- [Background] Sharma RK, Parashar A. Special considerations in paediatric burn patients. Indian J Plast Surg. 2010 Sep;43(Suppl):S43-50. doi: 10.4103/0970-0358.70719. PMID 21321657
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Pattanshetty RB, Gaude GS. Effect of multimodality chest physiotherapy in prevention of ventilator-associated pneumonia: A randomized clinical trial. Indian J Crit Care Med. 2010 Apr;14(2):70-6. doi: 10.4103/0972-5229.68218. PMID 20859490
- [Background] Cao Z. Application of Drainage Position Ventilation and Real-Time Bedside Monitoring in Mechanical Ventilation of Patients Infected with nCov-19. J Anaesth Ther. 2020;2(104):2.